CLINICAL TRIAL: NCT01440062
Title: Phase II Study of Efficacy of Vitamin D Supplementation in Multiple Sclerosis
Brief Title: Efficacy of Vitamin D Supplementation in Multiple Sclerosis (EVIDIMS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Jan-Markus Dörr, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EVIDIMS
Record Dates: First submitted 2011-09-19; First posted 2011-09-26 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum (high dose) (Experimental): verum arm receiving high dose Vitamin D oil
  Interventions: Drug: Verum arm receiving Vitamin D oil
- Verum (low dose) (Experimental): low dose arm receiving neutral oil and low dose of Vitamin D
  Interventions: Drug: low dose arm receiving neutral oil and 400 IU/g of Vitamin D every second day

INTERVENTIONS:
Drug: Verum arm receiving Vitamin D oil — oil: 20000 IU/g tablet: 400 IU/g every second day
  Arms: Verum (high dose)
Drug: low dose arm receiving neutral oil and 400 IU/g of Vitamin D every second day — neutral oil and a low dose of vitamin D
  Arms: Verum (low dose)

SUMMARY:
Examination of efficacy, safety and tolerability of vitamin D3 in the treatment of Multiple Sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age between 18 and 65 at randomization
* Relapsing-remitting MS according to the revised McDonald-Criteria (2005)
* EDSS ≤ 6,0
* Stable immunomodulatory treatment for at least 3 months
* Sufficient birth control (Pearl-Index <1) and negative pregnancy test at screening/randomization

Exclusion Criteria:

* Any other MS-course than RRMS
* Treatment with high dose vitamin D within 6 months prior to randomization
* Patients who have received over the last three months prior to randomization, an immunomodulatory therapy with the exception of IFN-β1b (Betaferon ®)
* Any condition that could interfere with MRI or other study related investigation
* Intolerability to Gd-DTPA
* Hypersensitivity to the drug Colecalciferol
* Patients with sarcoidosis
* Presence or history of nephrolithiasis
* Pseudohypoparathyroidism
* Clinically relevant dysfunction of liver, bone narrow or kidney defined by the following laboratory values:

  * HB <8.5 g / dl
  * WBC <2.5 / nl
  * platelet count <100/nl
  * Creatinine clearance by Cockcroft-Gault formula: Cl <110ml/min (male) and Cl <95ml/min (female)
  * AST / ALT> 3.5 times higher than the upper reference value
  * bilirubin> 2.0 mg / dl
  * hypercalcaemia> 2.7 mmol / l
  * calcium / creatinine ratio in urine> 1
* Treatment with hydrochlorothiazide, digitoxin, digoxin, phenytoin, barbiturates
* Pregnancy or lactation period
* Participation in any clinical study within 3 months before or at any time during study
* Any medical, psychiatric or other condition that could interfere with the patient's ability to understand and give the informed consent, to comply with the protocol or to finish the study any ruling commitment or placement in an institution

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Efficacy parameters | 1 day
  efficacy of Vitamin D (high dose) in patients with Multiple Sclerosis compared to low dose of Vitamin D

SECONDARY OUTCOMES:
Safety & tolerability parameters | 1 day
  Routine laboratory, vital signs, physical examination, ECG, AE reporting, Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Markus Dörr, Dr., Study Director — Charite; Jan-Markus Dörr, Dr., Principal Investigator — Charite-NeuroCure
Locations (6):
- Germany (6):
  - Kliniken für Neurologie Teupitz/Lübben, Asklepios Fachkliniken Brandenburg GmbH, Teupitz, Brandenburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Neurologische Praxis, Berlin
  - Neurologisches Facharztzentrum, Berlin
  - Krankenhaus Martha-Maria Halle-Dölau gGmbH, Halle
  - Sankt Josefs Krankenhaus Potsdam Neurologie, Potsdam

REFERENCES:
- [Derived] Backer-Koduah P, Infante-Duarte C, Ivaldi F, Uccelli A, Bellmann-Strobl J, Wernecke KD, Sy M, Demetriou M, Dorr J, Paul F, Ulrich Brandt A. Effect of vitamin D supplementation on N-glycan branching and cellular immunophenotypes in MS. Ann Clin Transl Neurol. 2020 Sep;7(9):1628-1641. doi: 10.1002/acn3.51148. Epub 2020 Aug 23. PMID 32830462
- [Derived] Dorr J, Backer-Koduah P, Wernecke KD, Becker E, Hoffmann F, Faiss J, Brockmeier B, Hoffmann O, Anvari K, Wuerfel J, Piper SK, Bellmann-Strobl J, Brandt AU, Paul F. High-dose vitamin D supplementation in multiple sclerosis - results from the randomized EVIDIMS (efficacy of vitamin D supplementation in multiple sclerosis) trial. Mult Scler J Exp Transl Clin. 2020 Jan 24;6(1):2055217320903474. doi: 10.1177/2055217320903474. eCollection 2020 Jan-Mar. PMID 32047645
- [Derived] Dorr J, Ohlraun S, Skarabis H, Paul F. Efficacy of vitamin D supplementation in multiple sclerosis (EVIDIMS Trial): study protocol for a randomized controlled trial. Trials. 2012 Feb 8;13:15. doi: 10.1186/1745-6215-13-15. PMID 22316314